CLINICAL TRIAL: NCT07162350
Title: Food as Medicine (FAME): An Innovative Approach to Improve Health and Nutrition Security Among High-Risk Children and Families in South Dallas
Brief Title: Food as Medicine Study
Acronym: FAME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parkland Health and Hospital System (Other)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jaclyn Albin, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU20251104
Record Dates: First submitted 2025-07-01; First posted 2025-09-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Chronic Diseases in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): The Usual Care control group reflects current clinical practices given to patients. This includes having access to routine wrap around services such as consultation with a dietitian and nutrition education materials. Providers provide references to applicable wrap around services; however, it is ultimately up to the patient to decide to utilize the resources.
- FAME (Experimental): The FAME intervention will be evaluated with a pragmatic randomized clinical trial. FAME will use a community health worker food navigator embedded in clinical settings to provide education and linkage to a community-based food hub that provides access to community driven food resources.
  Interventions: Behavioral: Food Navigation

INTERVENTIONS:
Behavioral: Food Navigation — For those randomized to the FAME Intervention, it will begin with a Community Health Worker (CHW) Food Navigator consultation. The role of the Food Navigators is as follows:
  1. Identify the top dietary and food needs of the participant and their family. The Food Navigator will perform a needs assessment to define food access, kitchen resources/capacity, and other social determinants of health.
  2. Set realistic, participant and family-driven nutrition goals. The Food Navigator will utilize Motivational Interviewing (MI), an evidence-based method of counseling that promotes motivation for change.
  3. Provide nutrition resources and referrals.
  4. Support children and families for up to 12 months.
  Arms: FAME

SUMMARY:
The Food as Medicine (FAME) intervention aims to improve dietary quality in lower income, primarily ethnic minority youth through food navigation that bridges clinical care and community food resources. This study will evaluate the FAME intervention on dietary quality, food behaviors, health outcomes, and cost-effectiveness, using a pragmatic randomized clinical trial design in 250 at risk youth (8-15 years of age) and their caregiver(s) as compared to Usual Care through the following aims:

Aim 1: To evaluate the impact of the FAME intervention on child and caregiver(s) dietary quality at 6 and 12 months as compared to Usual Care. Hypothesis: FAME participants will have increased dietary quality as measured by ASA-24/DQI.

Aim 2: To assess the intervention's impact on food behaviors, food insecurity, healthy food sourcing, knowledge, self-efficacy, health outcomes and cost-effectiveness at 6 and 12 months as compared to Usual Care.

Aim 3: Evaluate implementation outcomes including dose, satisfaction, and individual interviews and focus groups with youth, parents, physicians, clinic staff, community partners, and CHWs.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 8-15 years,
* BMI > 85th percentile, and
* be seen at one of the selected Parkland COPC (Community Oriented Primary Care) clinics.
* Both the participant and caregiver must be fluent in English or Spanish (read, write, and speak) and be willing to participate in the study over a 12-month duration.

Exclusion Criteria:

* has seen a dietitian within the last year,
* presence of an intellectual disability,
* diagnosed with autism with severe feeding difficulties,
* past medical history of severe feeding difficulties over the age of 2 years,
* has had bariatric surgery
* is taking a GLP-1
* diagnosed with type 1 diabetes
* is taking anti-psychotics
* has severe food allergies
* has a severe psychiatric disorder
* has a disease that would not allow the individual to change their diet, and
* any other reason the PIs deem someone ineligible.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Dietary Quality as measured by Diet Quality Index International (DQI-I) | Baseline to 6-months post-intervention
  Dietary quality is measured with the ASA 24-hour dietary recall (ASA 24) and the Diet Quality Index International (DQI-I). The ASA 24 is web-based tool that allows individuals to self-report all foods and beverages consumed in the previous 24 hours ((i.e., the data collection method). The DQI-I is a validated scoring system designed to assess overall diet quality (i.e., measure used to interpret the collected data). Used together, researchers will apply the DQI-I scoring algorithm to the nutrient and food group data collected from ASA 24 to generate a numeric DQI-I score that indicates the overall daily diet quality of the study participant. The DQI-I includes four components (variety 0-20; adequacy 0-40; moderation 0-30; overall balance 0-10) that contribute to a total score out of 100 points with higher scores indicating better diet quality. This allows us to track diet quality changes over time.

SECONDARY OUTCOMES:
Change in Dietary Quality as measured by Diet Quality Index International (DQI-I) | Baseline to 12-months post-intervention
  Dietary quality is measured with the ASA 24-hour dietary recall (ASA 24) and the Diet Quality Index International (DQI-I). The ASA 24 is web-based tool that allows individuals to self-report all foods and beverages consumed in the previous 24 hours ((i.e., the data collection method). The DQI-I is a validated scoring system designed to assess overall diet quality (i.e., measure used to interpret the collected data). Used together, researchers will apply the DQI-I scoring algorithm to the nutrient and food group data collected from ASA 24 to generate a numeric DQI-I score that indicates the overall daily diet quality of the study participant. The DQI-I includes four components (variety 0-20; adequacy 0-40; moderation 0-30; overall balance 0-10) that contribute to a total score out of 100 points with higher scores indicating better diet quality. This allows us to track diet quality changes over time.
Change in Resilience as measured by the Brief Resilience Scale (BRS) | Baseline to 6-months post-intervention
  The 6-item BRS uses a 5-point Likert scale (1 = strongly disagree, 2 = disagree, 3 = neutral, 4 = agree, 5 = strongly agree). Items 1, 3, and 5 are positively worded, and items 2, 4, and 6 are negatively worded. The BRS is scored by reverse coding items 2, 4, and 6 and finding the mean of the 6 items. A higher score indicates a higher level of resilience.
Change in Resilience as measured by the Brief Resilience Scale (BRS) | Baseline to 12-months post-intervention
  The 6-item BRS uses a 5-point Likert scale (1 = strongly disagree, 2 = disagree, 3 = neutral, 4 = agree, 5 = strongly agree). Items 1, 3, and 5 are positively worded, and items 2, 4, and 6 are negatively worded. The BRS is scored by reverse coding items 2, 4, and 6 and finding the mean of the 6 items. A higher score indicates a higher level of resilience.
Change in perceived stress as measured by the Perceived Stress Scale (PSS) | Baseline to 6-months post-intervention
  The 10-item PSS uses a 5-point Likert scale (0 = Never, 1 = Almost Never, 2 = Sometimes, 3 = Fairly Often, 4 = Very Often). PSS scores are obtained by reversing responses to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. Higher scores indicate higher levels of perceived stress.
Change in perceived stress as measured by the Perceived Stress Scale (PSS) | Baseline to 12-months post-intervention
  The 10-item PSS uses a 5-point Likert scale (0 = Never, 1 = Almost Never, 2 = Sometimes, 3 = Fairly Often, 4 = Very Often). PSS scores are obtained by reversing responses to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. Higher scores indicate higher levels of perceived stress.
Change in social support as measured by the Medical Outcomes Study (MOS) Social Support Survey | Baseline to 6-months post intervention
  The Medical Outcomes Study (MOS) Social Support Survey is a self-administered questionnaire that that includes 19 items across four functional support subscales: emotional/informational support (8 items), tangible/instrumental support (4 items), affectionate support (3 items), and positive social interaction (3 items). Each item is scored on a 5-point Likert style scale (1 = None of the Time; 5 = All of the Time) to indicate how often that type of support is available to them. A score for each social support subscale can be computed by averaging across the individual items or by adding scores individual items together. Higher scores indicate more support.
Change in social support as measured by the Medical Outcomes Study (MOS) Social Support Survey | Baseline to 12-months post intervention
  The Medical Outcomes Study (MOS) Social Support Survey is a self-administered questionnaire that that includes 19 items across four functional support subscales: emotional/informational support (8 items), tangible/instrumental support (4 items), affectionate support (3 items), and positive social interaction (3 items). Each item is scored on a 5-point Likert style scale (1 = None of the Time; 5 = All of the Time) to indicate how often that type of support is available to them. A score for each social support subscale can be computed by averaging across the individual items or by adding scores individual items together. Higher scores indicate more support.
Change in food security as measured by a standard measure from the USDA Economic Research Services | Baseline to 6-months post intervention
  The six-item standard measure from the U.S. Department of Agriculture (USDA) Economic Research Service is modeled using information from the Community Population Survey, Bureau of Labor Statistics, and American Community Survey. Food security status is assigned as follows: Raw score 0-1 - High or marginal food security (raw score 1 may be considered marginal food security, but a large proportion of households that would be measured as having marginal food security using the household or adult scale will have raw score zero on the six-item scale) Raw score 2-4 - Low food security Raw score 5-6 - Very low food security
Change in food security as measured by a standard measure from the USDA Economic Research Services | Baseline to 12-months post intervention
  The six-item standard measure from the U.S. Department of Agriculture Economic Research Service is modeled using information from the Community Population Survey, Bureau of Labor Statistics, and American Community Survey. Food security status is assigned as follows: Raw score 0-1 - High or marginal food security (raw score 1 may be considered marginal food security, but a large proportion of households that would be measured as having marginal food security using the household or adult scale will have raw score zero on the six-item scale) Raw score 2-4 - Low food security Raw score 5-6 - Very low food security
Change in parental self-efficacy as measured by the Parental Self-Efficacy for Healthy Dietary and Physical Activity Behaviors in Preschoolers Scale (PDAP) | Baseline to 6-months post intervention
  Parental self-efficacy (PSE) refers to beliefs of parents to effectively engage in behaviors that result in desired outcomes for their children. The PDAP instrument measures PSE in relation to contextual circumstances, for example, psychological states and situational demands. Responses are made according to an 11-point Likert scale, with anchors at 0 (not at all confident), 5 (moderately confident), and 10 (completely confident). A higher score indicates a higher level of PSE.
Change in parental self-efficacy as measured by the Parental Self-Efficacy for Healthy Dietary and Physical Activity Behaviors in Preschoolers Scale (PDAP) | Baseline to 12-months post intervention
  Parental self-efficacy (PSE) refers to beliefs of parents to effectively engage in behaviors that result in desired outcomes for their children. The PDAP instrument measures PSE in relation to contextual circumstances, for example, psychological states and situational demands. Responses are made according to an 11-point Likert scale, with anchors at 0 (not at all confident), 5 (moderately confident), and 10 (completely confident). A higher score indicates a higher level of PSE.
Change in child self-efficacy as measured by the Self-Efficacy to Regulate Eating Behaviors Scale for Children (SEREB-C) | Baseline to 6-months post intervention
  The SEREB-C is a 14-item self-report tool designed to measure children's perceived self-efficacy to choose healthy eating behaviors in challenging contexts. The points of the individual items are summed to create a composite score ranging from 8 to 40 for the activation and temptation situations subscale and from 6 to 30 for the negative emotional situations subscale (combined, total score ranges from 14 to 70). Higher scores imply greater self-efficacy in regulating eating behaviors in challenging situations.
Change in child self-efficacy as measured by the Self-Efficacy to Regulate Eating Behaviors Scale for Children (SEREB-C) | Baseline to 12-months post intervention
  The SEREB-C is a 14-item self-report tool designed to measure children's perceived self-efficacy to choose healthy eating behaviors in challenging contexts. The points of the individual items are summed to create a composite score ranging from 8 to 40 for the activation and temptation situations subscale and from 6 to 30 for the negative emotional situations subscale (combined, total score ranges from 14 to 70). Higher scores imply greater self-efficacy in regulating eating behaviors in challenging situations.
Change in dietary behavior as measured by the Mini-EAT survey | Baseline to 6-months post-intervention
  The Mini-EAT (Eating Assessment Tool) is a dietary assessment tool designed to evaluate the quality of a person's diet. It ranges from a low of 36 to a high of 90. Scores are categorized into three levels: unhealthy (<61), intermediate (61-69), and healthy (69<)
Change in dietary behavior as measured by the Mini-EAT survey | Baseline to 12-months post-intervention
  The Mini-EAT is a dietary assessment tool designed to evaluate the quality of a person's diet. It ranges from a low of 36 to a high of 90. Scores are categorized into three levels: unhealthy (<61), intermediate (61-69), and healthy (69<)
Change in BMI of child participants at 6 months post-intervention | Baseline to 6-months post-intervention
  Child health outcomes will be evaluated with electronic health records, including body mass index (BMI) (weight and height will be combined to report BMI in kg/m^2).
Change in BMI of child participants at 12 months post-intervention | Baseline to 12-months post-intervention
  Child health outcomes will be evaluated with electronic health records, including body mass index (BMI) (weight and height will be combined to report BMI in kg/m^2).
Change in Blood pressure of child participants at 6 months post-intervention | Baseline to 6-months post-intervention
  Child health outcomes will be evaluated with electronic health records, including systolic and diastolic blood pressure data.
Change in Blood pressure of child participants at 12 months post-intervention | Baseline to 12-months post-intervention
  Child health outcomes will be evaluated with electronic health records, including systolic and diastolic blood pressure data.
Change in Glycated hemoglobin (HbA1c) of child participants at 6 months post-intervention | Baseline to 6-months post-intervention
  Child health outcomes will be evaluated with electronic health records, including glycated hemoglobin (HbA1c) data.
Change in Glycated hemoglobin (HbA1c) of child participants at 12 months post-intervention | Baseline to 12-months post-intervention
  Child health outcomes will be evaluated with electronic health records, including glycated hemoglobin (HbA1c) data.
Change in Alanine transaminase (ALT) of child participants at 6 months post-intervention | Baseline to 6-months post-intervention
  Child health outcomes will be evaluated with electronic health records, including alanine transaminase (ALT) data.
Change in Alanine transaminase (ALT) of child participants at 12 months post-intervention | Baseline to 12-months post-intervention
  Child health outcomes will be evaluated with electronic health records, including alanine transaminase (ALT) data.

CONTACTS AND LOCATIONS:
Overall Officials: Jaclyn Albin, MD, Principal Investigator — Parkland Health
Locations (1):
- Parkland Health & Hospital System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share individual participant data (IPD) with other researchers. If this decision changes, an IPD sharing plan will be provided according to institutional regulations at a later time.